CLINICAL TRIAL: NCT07066085
Title: Serial Blood Count Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, David Dale, Professor, Division of Internal Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00020909
Record Dates: First submitted 2025-06-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cyclic Neutropenia; Congenital Neutropenia; Neutropenia
Keywords: Neutropenia; Cyclic Neutropenia; Congenital Neutropenia; Device
MeSH Terms: conditions — Cyclic neutropenia; Neutropenia, Severe Congenital, Autosomal Recessive 3; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Serial Blood Count Study (Experimental)
  Interventions: Device: Serial Blood Count Study; Device: Athelas Home device

INTERVENTIONS:
Device: Serial Blood Count Study — A new home monitoring device called Athelas One (or Athelas Home) was granted an FDA 510K Class 2 clearance for evaluation of white blood count (WBC) and absolute neutrophil count (ANC).
  The device uses a drop of blood on a slide to measure the WBC and ANC. The drop of blood is obtained using a lancet that comes with the device, it is just like how diabetics do with a glucose monitoring device. The process will be done once a day for 42 days (6 weeks) unless the drop is not placed on the slide correctly. If there is an issue with the first attempt, the process could be done again to obtain the WBC and ANC results.
  The Athelas device is intended for use by patients with neutropenia or patients at risk of neutropenia. The device is indicated for use by patients and caregivers within home settings with results viewable by health care professionals.
Device: Athelas Home device — A new home monitoring device called Athelas One (or Athelas Home) was granted an FDA 510K Class 2 clearance for evaluation of white blood count (WBC) and absolute neutrophil count (ANC).
  The device uses a drop of blood on a slide to measure the WBC and ANC. The drop of blood is obtained using a lancet that comes with the device, it is just like how diabetics do with a glucose monitoring device. The process will be done once a day for 42 days (6 weeks) unless the drop is not placed on the slide correctly. If there is an issue with the first attempt, the process could be done again to obtain the WBC and ANC results.
  The Athelas device is intended for use by patients with neutropenia or patients at risk of neutropenia. The device is indicated for use by patients and caregivers within home settings with results viewable by health care professionals.

SUMMARY:
The objective of the Serial Blood Count Study is to determine the utility of home monitoring of white blood cell (WBC) and absolute neutrophil counts (ANC) to diagnose cyclic neutropenia and distinguish between cyclic and severe congenital neutropenia (SCN). A new home monitoring device called Athelas One was granted an FDA 510K Class 2 clearance for evaluation of white blood count (WBC) and absolute neutrophil count (ANC). The investigators believe this device provides a unique and extremely valuable opportunity to for diagnosis of these diseases.

DETAILED DESCRIPTION:
The objective of the Serial Blood Count Study is to determine the utility of home monitoring of white blood cell (WBC) and absolute neutrophil counts (ANC) to diagnose cyclic neutropenia and distinguish between cyclic and severe congenital neutropenia (SCN). A new home monitoring device called Athelas One was granted an FDA 510K Class 2 clearance for evaluation of white blood count (WBC) and absolute neutrophil count (ANC). The investigators believe this device provides a unique and extremely valuable opportunity to for diagnosis of these diseases.

Cyclic neutropenia (CyN) usually occurs as an autosomal dominant disorder caused by mutations in the gene for neutrophil elastase, ELANE. Severe congenital neutropenia (SCN) is also hereditary and caused by mutations in the same gene. Distinguishing between these diseases by genotyping is imprecise because of overlap in the mutational profiles. However, the distinction is critical because SCN has a far greater risk of evolution to myelodysplasia (MDS) and acute myeloid leukemia (AML). The risk is approximately 20-25% for patients with SCN and less than 1% for CyN. Because of this risk, patients with SCN are likely to be referred for hematopoietic stem cell transplantation (HSCT), whereas CyN patients are not. The best way to distinguish between these conditions is with serial ANC determinations. It is not easy for subjects to get 6 weeks of daily blood counts because this requires repeated trips to a clinical laboratory for blood draws, usually from a vein in the arm. From the subject's and family's perspective, the trips are time-consuming and expensive, testing is expensive, and the blood draws often lead to bruising and arm pain from repeated pokes. The goal of the study is to learn if patients will be compliant with use of the fingerstick technique to obtain a blood sample for 6 weeks and see the results of the WBC and ANC results so that clinicians can clearly distinguish between the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of severe chronic neutropenia
* 5 years of age or older, male or female
* Known positive ELANE mutation
* Computer if available
* Internet access
* Cell phone / Smart phone that can download / install applications (App)
* Adults that are comfortable obtaining the samples without medical conditions that would make collection of the sample difficult.

Exclusion Criteria:

* Diagnosis of severe chronic neutropenia and negative results for the ELANE mutation
* Less than 5 years of age
* No internet access
* No Cell phone or smart phone that cannot download / install applications (App)
* Adults that are uncomfortable obtaining the samples or have medical conditions that would make collection of the sample difficult.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Test feasibility of device for white blood cell (WBC) count | Daily blood counts over a period of 42 days (6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Dale, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center - Montlake, Seattle, Washington, United States